CLINICAL TRIAL: NCT02279628
Title: Continuous Pre-uterine Wound Infiltration Versus Intrathecal Morphine for Postoperative Analgesia After Cesarean Section. Controlled Comparative Study.
Brief Title: Continuous Pre-uterine Wound Infiltration Versus Intrathecal Morphine for Postoperative Analgesia After Cesarean Section
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Maternite Regionale Universitaire (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012-004498-14
Record Dates: First submitted 2014-10-16; First posted 2014-10-31 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Postoperative Pain
Keywords: cesarean section; spinal anesthesia; continuous wound infiltration; intrathecal morphine; oral morphine
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Continuous wound infiltration alone (Experimental): Spinal anesthesia will be performed with 10 mg bupivacain 0.5% hyperbaric, 3 μg sufentanil and 1 ml sodium chloride 0.9% (without morphine). Patient will then receive a continuous wound infiltration of ropivacaine 0.2% 8 ml/H via a preperitoneal catheter.
  Interventions: Drug: Ropivacaine
- Intrathecal moprhine alone (Active Comparator): Spinal anesthesia will be performed with 10 mg bupivacain 0.5% hyperbaric, 3 μg sufentanil and 0.1mg morphine. Patient will then receive a continuous wound infiltration of sodium chloride 0.9% 8 ml/H via a preperitoneal catheter.
  Interventions: Drug: Morphine
- Intrathecal morphine&wound infiltration (Experimental): Spinal anesthesia will be performed with 10 mg bupivacain 0.5% hyperbaric, 3 μg sufentanil and 0.1mg morphine. Patient will then receive a continuous wound infiltration of ropivacaine 0.2% 8 ml/H via a preperitoneal catheter.
  Interventions: Drug: Ropivacaine; Drug: Morphine

INTERVENTIONS:
Drug: Ropivacaine — Ropivicaine (0.2%) bolus of 10ml will be injected through the catheter after surgery and continuously infused during the postoperative period (8ml/H)
  Arms: Continuous wound infiltration alone; Intrathecal morphine&wound infiltration
Drug: Morphine — Morphine will be injected intrathecally (100µg) and oral morphine will be given during the postoperative period
  Arms: Intrathecal moprhine alone; Intrathecal morphine&wound infiltration

SUMMARY:
The cesarean section is considered as a painful surgery during the post operative period. Mothers may need to move immediately after the surgery to take care of their babies. This may increase the risk of major pain and chronic pain. Thus, excellent postoperative analgesia is required so that mothers do not experience pain in caring for their baby. Currently, several techniques have been developed to manage postoperative pain related to c-section scar such as intrathecal morphine during spinal anesthesia or continuous pre-peritoneal wound infiltration. The comparison between anesthetic techniques has never been performed and it is still not know if the combination of intrathecal morphine plus continuous pre-peritoneal wound infiltration provide a synergistic or additional effect on pain relief.

DETAILED DESCRIPTION:
The aim of this study is to compare the efficacy of continuous wound infiltration versus intrathecal morphine for postoperative analgesia after scheduled cesarean section. The primary endpoint is morphine consumption during the first 48 postoperative hours.

ELIGIBILITY:
Inclusion Criteria:

* Elective Cesarean section
* Spinal anesthesia
* Singleton
* ASA ( Physical status score) 1 to 3

Exclusion Criteria:

* Age <18yrs
* BMI ≥ 45 kg/m2 or weight < 45 kg
* Refusal to consent
* Urgent cesarean section
* Allergy to a medication used in the protocol
* Impaired hemostasis ou current infection
* Contra indication or failure of spinal anesthesia

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Morphine consumption during the first 48 postoperative hours | at the 48th hour

SECONDARY OUTCOMES:
Pain at rest and at mobilization | Every 4 hours during the first 48 postoperative hours
  The pain at rest and at mobilization will be evaluated with both Visual Analog scale and Verbal pain scale. The patient should describe the worst pain felt during the previous 4 hours in a lying position and at mobilization
Time to restoration of bowel function | within the first 48 postoperative hours
Verbal and Visual analog pain scores in the first standing position | at day 1
Number of patients that required oral morphine | At the 24th and 48th hour
Number of patients that required local anesthetic rescue dose through the catheter | At the 24th and 48th hour
Postoperative rehabilitation survey | At the 48th hour
Occurrence of side effect | During the first 48 hours
  Itching, nausea and vomiting, drowsiness, urinary retention, hypoventilation, other will be assessed with a questionnaire
Postoperative residual pain (DN4 survey) | At 3 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Hervé BOUAZIZ, MD., PhD., Study Chair — Department of Anesthesiology, Maternité Régionale Universitaire, CHU NANCY, France; Florence VIAL, MD., Principal Investigator — Department of Anesthesiology, Maternité Régionale Universitaire, CHU NANCY, France; Philippe GUERCI, MD, Principal Investigator — Department of Anesthesiology and Critical Care Medicine, CHU NANCY Brabois, FRANCE
Locations (1):
- Maternité Régionale Universitaire (MRU), Nancy, Lorraine, France

REFERENCES:
- [Derived] Viviand C, Pietretti E, Luc A, Herbain D, Baka N, Morel O, Feugeas J, Aron C, Bouaziz H, Guerci P, Vial F. Continuous wound infusion combined with intrathecal morphine for analgesia after Cesarean delivery compared with intrathecal morphine or continuous wound infusion alone. Can J Anaesth. 2022 Jun;69(6):788-789. doi: 10.1007/s12630-022-02223-2. Epub 2022 Mar 10. PMID 35274209